CLINICAL TRIAL: NCT03001752
Title: Evaluation of Morphological and Dimensional Alveolar Bone Changes Around Post-extraction Implants in an Open Flap, Open Flap and Grafting and Flapless Technique. A Clinical Randomized Controlled Study
Brief Title: Immediate Implants Inserted Through Open Flap, Open Flap and Bone Grafting and Flapless Techniques
Acronym: ETPEI-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Felice Roberto Grassi, Professor, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4987
Record Dates: First submitted 2016-12-16; First posted 2016-12-23 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Isolated Premolar Edentulous Site
Keywords: post-extraction dental implant; immediate dental implant; open flap; flapless; bone grafting; CT Cone Beam
MeSH Terms: interventions — Dental Implants; Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The care provider could not be blinded because of the nature of the treatment. The patient was blinded and the investigator and outcome assessor as well (using a code to identify teeth and patients).
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open flap immediate implant (Active Comparator): Open flap immediate implant insertion, without bone grafting
  Interventions: Device: Open flap immediate implant
- Open flap immediate implant and bone grafting (Active Comparator): Open flap immediate implant insertion and bone grafting
  Interventions: Device: Open flap immediate implant and bone grafting
- Flapless immediate implant (Active Comparator): Immediate implant insertion without opening flap of inserting bone grafting
  Interventions: Device: Flapless immediate implant

INTERVENTIONS:
Device: Open flap immediate implant — Post-extraction implants will be inserted through open flap, without bone grafting
  Other Names: Dental implant
  Arms: Open flap immediate implant
Device: Open flap immediate implant and bone grafting — Post-extraction implants will be inserted through open flap, adding bone grafting
  Other Names: Dental implant, bone grafting
  Arms: Open flap immediate implant and bone grafting
Device: Flapless immediate implant — Post-extraction implants will be inserted without elevating flap or inserting bone grafting
  Arms: Flapless immediate implant

SUMMARY:
This is a three-armed randomized controlled clinical trial aiming the estimation of dimensional alveolar bone changes after insertion of post-extraction implants through 3 different surgical techniques: open flap, open flap and grafting, flapless.

DETAILED DESCRIPTION:
Background and Objectives A recent systematic review investigating dimensional alveolar bone changes after insertion of post-extraction implants reported that there is a lack of randomized controlled trials that would serve as a scientific base for building clinical guidelines on alveolar site treatment after insertion of post-extraction implants. Different studies suggest that insertion of post-extraction implants should be performed after fully elevating a flap and inserting bone graft in the residual space between the implant surface and the alveolar socket. Other investigations report insignificant differences between open flap and flapless approaches, whereas the insertion of bone grafts remains controversial.

The present study is a three-armed randomized clinical controlled trial conducted with the following objectives:

1. Evaluation of morphological and alveolar bone level differences (marginal bone loss) on post-extraction implants inserted with the following techniques: 1) open flap surgery alone; 2) open flap surgery and bone grafting; 3) flapless.
2. Estimation of effectiveness of the three surgical techniques through measurement of secondary outcomes such as intra-operatory and post-operatory complications, pain and discomfort, time and costs.

Materials and Methods

* This is a three-armed randomized controlled clinical trial where each arm will belong to one of the treatments: 1) open flap surgery alone; 2) open flap surgery and bone grafting; 3) flapless.
* The randomizing sequence will be generated from a computer program (STATA 13) by a statistician who will also conduct blind statistical analysis of results.
* All patients will be recruited prior to trial commencement. They will be extensively informed regarding the intervention and will sign a treatment consent.
* Patients will be recruited according to the following inclusion criteria: absence of any systemic disease that might compromise implant integration or wound healing, appropriate periodontal health (measured through periodontal indexes), presence of premolars with indications of extractions, presence of adjacent teeth, absence of fenestrations, presence of vestibular alveolar wall with a minimum of 0.5mm of thickness. Patients who have undergone CT scanning in the past 5 years and heavy smokers (more than 20 cigarettes per day) will not be included in the study.
* Calculation of sample size has already been performed by an experienced statistician, accounting for a minimal predicted difference between groups of 1mm (SD 0.75mm) of marginal bone loss, alpha error of 0.05 and 90% of power. Based on these calculations, a total of 45 patients will be included in the study.
* Interventions will be performed in accordance with ethical standards as suggested by the Helsinki Declaration (1975). Approval of Ethical Committee of the University of Bari has already been obtained (reg.nr. 4987).
* All surgical interventions will be performed by the same experienced surgeon who will be informed of the type of intervention after tooth extraction (allocation concealment through dark sealed envelopes).
* The primary outcome is marginal bone loss (MBL) and alveolar bone dimensional changes measured through CT Cone Beam performed immediately after implant insertion and 6 months after. Secondary outcomes are intra-and post-operative complications, pain and discomfort, time and costs.
* Outcomes will be measured by another clinician blinded in terms of treatment allocation.
* Statistical analysis will be performed by an independent statistician. Statistical tests will include: One-way Anova, Bonferroni tests and several linear and logistic regressions in order to estimate potential predictive variables. Statistical significance will be set at .05.
* Interruption of study will be considered in the following situations: 1.preliminary observation of highly significant difference between techniques indicating one technique highly superior; 2. big number of lost to follow-up (bigger than that considered during sample size calculation)
* Patients will be excluded from the study in the following cases: missing follow-up hygiene controls at 1 and 3 months post-intervention, missing 6 months follow-up control, poor cooperation in terms of domestic oral hygiene (periodontal indexes measured), income of systemic or local diseases that might compromise outcomes.

ELIGIBILITY:
Inclusion Criteria:

* absence of any systemic disease that might compromise implant integration or wound healing
* appropriate periodontal health (measured through periodontal indexes)
* presence of premolars with indications of extractions, presence of adjacent teeth
* absence of fenestrations
* presence of vestibular alveolar wall with a minimum of 0.5mm of thickness

Exclusion Criteria:

* patients who have undergone CT scanning in the past 5 years
* heavy smokers (more than 20 cigarettes per day)
* patients not showing up at 1 and 3 months hygiene sessions
* patients not showing up at 6 months follow-up

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Marginal Bone Loss measured through CT Cone Beam | 6 months
  Difference of marginal bone level measured immediately after treatment and 6 months after on two repeated (immediately after and 6 months after implant insertion) CT Cone Beam
Alveolar Bone Dimensional Reduction assessed through CT Cone Beam | 6 months
  Three-dimensional Alveolar Bone Reduction (horizontal and vertical) will be measured on two repeated (immediately after and 6 months after implant insertion) on CT Cone Beam, having as reference points the implant platform and the implant apex.

SECONDARY OUTCOMES:
Pain and Discomfort measured through questionaire | 1 Week
  Pain and discomfort experienced by the patient after the surgery, measured through a VAS scale on a questionaire
Intra-operatory or post-operatory complications assessed through intra-operatory observation and post-intervention check-ups. | 6 months
  Intra-operatory or post-operatory intervention-related adverse events such as excessive bleeding, swallowing, hematoma will be recorded for each patient.
Time needed to perform surgical intervention | 1-2 hours
  Time needed to perform surgical intervention (immediately after tooth extraction until finishing of surgical procedure) will be recorded for each intervention.

REFERENCES:
- [Result] Lee CT, Chiu TS, Chuang SK, Tarnow D, Stoupel J. Alterations of the bone dimension following immediate implant placement into extraction socket: systematic review and meta-analysis. J Clin Periodontol. 2014 Sep;41(9):914-26. doi: 10.1111/jcpe.12276. Epub 2014 Jul 23. PMID 24894299
- [Result] Tarnow DP, Chu SJ. Human histologic verification of osseointegration of an immediate implant placed into a fresh extraction socket with excessive gap distance without primary flap closure, graft, or membrane: a case report. Int J Periodontics Restorative Dent. 2011 Sep-Oct;31(5):515-21. PMID 21845246